CLINICAL TRIAL: NCT05476939
Title: Biological Medicine for Diffuse Intrinsic Pontine Glioma (DIPG) Eradication
Brief Title: Biological Medicine for Diffuse Intrinsic Pontine Glioma (DIPG) Eradication 2.0
Acronym: BIOMEDE 2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Innovative Therapies For Children with Cancer Consortium (Other); Ministry of Health, France (Other Government); Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014/2126; 2014-001929-32 (EudraCT Number); 2023-506027-29-00 (EU CTIS Number)
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Diffuse Midline Glioma, H3 K27M-Mutant; Diffuse Midline Glioma, H3K27-altered
Keywords: Children; Adolescents; Adults; Newly diagnosed
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma | interventions — Everolimus; TIC10 compound; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- everolimus (Active Comparator): Tablets of 2.5 mg or 10 mg. The prescribed dose is 5 mg/m²/day, orally, once daily. Dose will be capped at 10 mg once daily.
  Treatment will be continued until unacceptable toxicity, centrally confirmed tumor progression (either radiologically or histologically) and/or withdrawal of patient, parents or legal representative consent.
  At the time of centrally confirmed relapse or progression, patients will stop treatment and will be allowed to switch to the other arm in case no better option is available after considering the results of the molecular profiling. In case of switch (everolimus to ONC201 or vice-versa), the patient will observe a wash-out period of 7 days before starting:
  * the second treatment,
  * or a reirradiation (if applicable). No treatment is allowed during reirradiation, except setroids and bevacizumab. Then, if an additional treatment is needed, the second treatment will be started within one week after the end of the reirradiation.
  Interventions: Drug: Everolimus; Radiation: Radiotherapy
- Dordaviprone (ONC201) (Experimental): Capsules of 125 mg. The prescribed dose is 375 mg/m², orally, once daily at Day 1 and Day 2 of each week.
  Dose will be capped at 625 mg per dose.
  Treatment will be continued until unacceptable toxicity, centrally confirmed tumor progression (either radiologically or histologically), and/or withdrawal of patient, parents or legal representative consent.
  At the time of centrally confirmed relapse or progression, patients will stop treatment and will be allowed to switch to the other arm in case no better option is available after considering the results of the molecular profiling. In case of switch (everolimus to ONC201 or vice-versa), the patient will observe a wash-out period of 7 days before starting:
  * the second treatment,
  * or a reirradiation (if applicable). No treatment is allowed during reirradiation, except setroids and bevacizumab. Then, if an additional treatment is needed, the second treatment will be started within one week after the end of the reirradiation.
  Interventions: Drug: ONC201; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Everolimus — Tablets of 2.5 mg or 10 mg. The prescribed dose is 5 mg/m²/day, orally, once daily. Dose will be capped at 10 mg once daily.
  Other Names: VOTUBIA; AFINITOR
  Arms: everolimus
Drug: ONC201 — Capsules of 125mg. The prescribed dose is 375mg/m², orally, once daily at Day 1 and Day 2 of each week.
  Dose will be capped at 625 mg per dose.
  Arms: Dordaviprone (ONC201)
Radiation: Radiotherapy — All patients will be treated with 30 conventional single daily fractions of 1.8 Gy to a total of 54 Gy over a planned period of 6 weeks. Dose may be increased up to 60 Gy for adult patients with supratentorial ND-DMG. The clinical target volume will include all the areas of abnormality on T2/FLAIR sequences with a 1-cm margin.
  Radiotherapy will have to start within a maximum of 4 weeks for DIPG, up to 6 weeks for other DMG H3K28-altered (ND-DMG), after the biopsy or last surgery. The study medication will be started at Day 1 (+3 days max) of radiotherapy. Reirradiation is permitted only at disease progression according to local practice.
  In case of metastatic disease or intramedullary tumors, patients can be included in the study. In this situation, radiotherapy will have to start within a maximum of 4 weeks for DIPG, up to 6 weeks for other DMG H3K28-altered (ND-DMG), after the biopsy or last surgery while targeted treatment will start at the end of the irradiation.

SUMMARY:
The BIOMEDE 2.0 study is the second stage of the BIOMEDE multi-arm, multistage rolling programme (adaptive platform protocol).

It is a multicenter, randomized, open-label, controlled phase-3 trial evaluating efficacy of ONC201 in comparison with everolimus (primary objective based on internal comparison) and subsequently to historical controls.

Two treatment groups will be compared. A switch between treatment groups is allowed after confirmation of the disease progression (real-time central review blinded to the treatment arm allocation). Study treatment will be continued until centrally confirmed disease progression (either radiologically or histologically), unacceptable toxicity or consent withdrawal.

The final conclusion of the trial will be successful for ONC201, if ONC201 is found significantly superior to everolimus in terms of centrally-reviewed PFS (Progression-free survival) from randomization (internal comparison) either overall, considering ND-DMG and DIPG-patients together, or in the subgroup of ND-DMG patients alone. In other cases, Everolimus will remain the standard arm unless it appears associated with an excess of toxicity compared to ONC201 which could then be discussed as a new standard.

ELIGIBILITY:
Eligibility criteria for the inclusion (registration) in BIOMEDE 2.0 study:

* Diagnosis Criteria:

  * Diagnosis of DIPG (clinical and radiological). As biopsy is not standard for these tumors, an informed consent is required for the necessary histological verification. [Biopsy-part of BIOMEDE 2.0 trial]. OR
  * Histological diagnosis of DIPG (i.e. H3K28M or EZHIP positive Diffuse Midline Glioma located in the pons) in case the tumor biopsy was performed before study entry. The diagnosis will be defined by 1/ diffuse glioma, 2/ H3K28M mutation or loss of H3K28 trimethylation together with EZHIP overexpression. In this situation, patient will sign the consent after the diagnosis to allow central review and biomarkers assessment thereafter. OR
  * Molecular diagnosis of DIPG (i.e. H3K28M) in case a liquid biopsy (CSF or blood) was performed before study entry, in a patient who could not undergo a tumor biopsy because it was too dangerous according to the patient's clinical condition. The diagnosis will be defined by 1/ DIPG, 2/ H3K28M mutation. In this situation, patient will sign the consent after the diagnosis to allow collection of the molecular report. OR
  * Non-DIPG diffuse midline gliomas (ND-DMG), H3K28M mutant or with H3K28 trimethylation loss together with EZHIP overexpression, will be eligible for the trial after biopsy or surgery. As biopsy and surgery is considered as standard practice for these locations, informed consent for the biopsy will not be necessary. Patient will sign the consent after the diagnosis to allow central review and biomarkers assessment thereafter. OR
  * Non-DIPG diffuse midline gliomas (ND-DMG) will be eligible for the trial before the biopsy in case the diagnosis is clinically or radiologically suspected. Informed consent for the biopsy and molecular analysis will be necessary. Then, if the central pathology review concludes to a ND-DMG with H3K28M mutant or H3K28 trimethylation loss together with EZHIP overexpression, these patients will be eligible for the treatment part of the trial.
* Eligible for a biopsy, or biopsy material available for the biomarker assessment.
* Age > 6 months, with no upper age limit. Children between 6 months and 3 years will be discussed on a case by case basis for inclusion in the study for the feasibility of the stereotactic biopsy.
* Eligible for cerebral or craniospinal radiotherapy.
* Tumor at diagnosis: no prior chemotherapy for the present cancer; no prior cerebral radiation therapy even for another neoplasm. Surgery is allowed when performed for diagnostic or therapeutic purpose.
* Metastatic diseases or spinal tumors allowed; in this case, patients would receive craniospinal or spinal radiotherapy and medical treatment (everolimus or ONC201) will be postponed and only started after the end of radiotherapy.
* Patients must be affiliated to a social security system or beneficiary of the same according to local requirements.
* Written informed consent from parents/legal representative, patient, and age-appropriate assent before any study-specific procedures are conducted according to local, regional or national guidelines.

Non eligibility criteria for the inclusion (registration) in BIOMEDE 2.0 study:

* Uncontrolled spontaneous massive intratumor bleeding. Patients with post-operative bleeding will be allowed to enter the study provided the hemorrhage is controled. Same rule applies for the other post-operative complications (infection, CSF leakage, absence of wound closure, subdural collection…).
* Any other concomitant anti-cancer treatment not foreseen by this protocol is not allowed, except corticosteroids and Bevacizumab which are allowed during the protocol. Bevacizumab is not allowed before and until 15 days after the surgery. The use of bevacizumab and corticosteroids will be taken into account when judging the possibility of progression/pseudoprogression.
* Any other cancer diagnosed during the last 5 years.
* Uncontrolled intercurrent illness or active infection.
* Any other co-morbid condition that in the investigator's opinion would impair study participation.
* Unable for medical follow-up (geographic, social or mental reasons).
* Patient previously treated with irradiation on the brainstem for another neoplasm.
* Participation in another clinical study with an investigational product while on study treatment.
* Patient under guardianship or deprived of his/her liberty by a judicial or administrative decision or incapable of giving his/her consent.

Eligibility criteria for the randomization in BIOMEDE 2.0 study:

* Patient enrolled in the BIOMEDE 2.0 study.
* Life expectancy > 12 weeks after the start of study treatment.
* Histological diagnosis of DIPG (as per the WHO criteria) confirmed by central pathology review, OR Typical radiology of a DIPG (mandatory central radiological review) as well as the short clinical history (less than three months of pre-existing symptoms) in case of suspected DIPG but no histological confirmation (tumor biopsy performed but not informative), or suspected DIPG with detection of H3K28M mutation in the CSF or blood (ctDNA analysis in the CSF or blood), OR Histological diagnosis of ND-DMG confirmed by central pathology review, with mutation in the histone H3.1, H3.2, H3.3 genes, or loss of H3K28me3 and EZHIP overexpression by immunohistochemistry.
* Karnofsky performance status scale or Lansky Play Scale > 50%. The PS should not take the neurologic deficit per se into account. NB: Children and adults with a worse performance status due to glioma-related motor paresis can be included.
* Highly effective and appropriate contraception for patients (male and female) of reproductive potential during their entire participation in the study and during 6 months after the end of treatment.
* Negative pregnancy test (serum beta-HCG or urinary test) evaluated within one week prior randomization in sexually active females of reproductive potential.
* Absolute neutrophil count > 1.0 x 10^9/l, Platelets > 100 x 10^9/l.
* Total bilirubin < 1.5 x ULN, AST and ALT< 2.5 x ULN.
* Serum creatinine < 1.5 X ULN for age. If serum creatinine > 1.5 x ULN, creatinine clearance must be > 70 ml/min/1.73 m² (as per local practice).
* Normal coagulation tests within the local reference ranges.
* Written informed consent from parents/legal representative, patient, and age-appropriate assent before randomization according to local, regional or national guidelines.

Non Eligibility criteria for the randomization in BIOMEDE 2.0 study:

* Current organ toxicity > grade 2 according to the NCI-CTCAE version 5.0, especially cardiovascular or renal disease (including but not limited to: congenital long QT syndrome, nephrotic syndrome, glomerulopathy, uncontrolled high blood pressure despite adequate treatment).
* Patients with the following cardiac history cannot take ONC201:

  * Prolongation of QT/QTcF interval (QTc interval > 480 milliseconds) preferably using Frederica's QT correction formula on two ECGs separated by at least 48 hours.
  * A history of Torsades de pointes or heart failure, hypokalemia, or family history of prolonged QT Syndrome.
  * Required concomitant use of medication(s) known to prolong the QT/QTc interval.

In this case, patients will be treated in the Everolimus arm without randomization (except if contra-indication to Everolimus).

* Pregnant or breastfeeding women.
* Patients with chronic HBV disease compatible with the trial are not excluded from the study. These patients randomized to everolimus treatment will have regular viral load monitoring throughout the study.
* Patients taking strong P450 inhibitors or inducers or PgP inhibitors are not excluded from the study but drug concentration of everolimus should be monitored carefully to avoid toxicity. Preferably alternative medications should be considered.
* Patient with known congenital galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption will not be randomized and will be treated in the ONC201 arm (except if contra-indication to ONC201).
* Patients with known hypersensitivity to any component of Everolimus (active substance, other rapamycin derivatives or excipients) will not be randomized and will be treated in the ONC201 arm (except if contra-indication to ONC201).
* Patients with known hypersensitivity to any component of ONC201 (drug product or excipients) will not be randomized and will be treated in the Everolimus arm (except if contra-indication to Everolimus).

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 433 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Until 2 years after inclusion of the last patient
  Defined as the time between date of randomization and unequivocal clinical, cytological or radiological progression confirmed by central review, or death whatever the cause.

SECONDARY OUTCOMES:
Overall survival (for all the comparisons to historical controls) | Until 5 years after randomization of the last patient
  Defined from the date of radiological diagnosis to the date of death from any cause.
Overall survival (for the internal comparison between randomized groups) | Until 5 years after randomization of the last patient
  Defined from the date of randomization to the date of death from any cause.
Progression-free survival after first progression | Until 5 years after randomization of the last patient
  It will also be computed from the date of progression to the date of subsequent progression or death from any cause, in order to describe the outcome after progression.
Complication rate of the diagnostic biopsy-based procedure | Until 5 years after randomization of the last patient
Severity of the complications (including prolongation of the hospital stay) of the diagnostic biopsy-based procedure | Until 5 years after randomization of the last patient
Duration of the complications (including delay for starting treatment) of the diagnostic biopsy-base procedure | Until 5 years after randomization of the last patient
Safety profile of the drugs | Until 5 years after randomization of the last patient
  Using the NCI-CTC v5.0 criteria, during radiotherapy and during the entire duration of the administration of the drug, considering all adverse events except adverse events unequivocally related to the disease (pseudo)-progression.
Relative benefit/risk ratio of ONC201 compared to everolimus | Until 5 years after randomization of the last patient
  It will be assessed using the Q-TWiST approach (Quality-adjusted time without symptoms of disease or adverse event) evaluated from survival times (overall survival and progression-free survival) and adverse events data (date of occurrence of grade 3+ adverse event).

CONTACTS AND LOCATIONS:
Overall Officials: Jacques GRILL, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (50):
- Denmark (3):
  - Aarhus Universitetshospital Skejby, Aarhus
  - Rigshospitalet, Copenhagen
  - H.C. Andersen Children's Hospital, Odense Universitetshospital, Odense
- France (43):
  - Gustave Roussy, Villejuif, Val de Marne
  - CHU d'Amiens-Picardie Site Sud, Amiens
  - Institut de Cancérologie de l'Ouest (ICO) - Site Paul Papin, Angers
  - CHU d'Angers - Bâtiment Robert Debré, Angers
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - CHU de Bordeaux - Groupe hospitalier Saint André - Hôpital Saint André, Bordeaux
  - CHU de Bordeaux - Groupe hospitalier Pellegrin - Hôpital des enfants, Bordeaux
  - CHRU de Brest - Hôpital Morvan, Brest
  - CHU de Caen - Hôpital Côte de Nacre, Caen
  - CHU Estaing, Clermont-Ferrand
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU François Mitterrand, Dijon
  - CHU Grenoble Alpes - Hôpital Albert Michallon, Grenoble
  - CHU Grenoble Alpes - Hôpital Couple-Enfant, Grenoble
  - Centre Oscar Lambret, Lille
  - Hôpital Roger Salengro, Lille
  - Hôpital de la mère et de l'enfant, Limoges
  - Centre Léon Bérard, Lyon
  - Hôpital Pierre Wertheimer, Lyon
  - Hôpital de La Timone, Marseille
  - Hôpital Arnaud de Villeneuve, Montpellier
  - CHRU Nancy - Hôpital central, Nancy
  - CHRU Nancy Brabois - Hôpital d'enfants, Nancy
  - CHU de Nice - Hôpital Pasteur 2, Nice
  - CHU de Nice - Hôpital L'Archet 2, Nice
  - Hôpital Saint Louis, Paris
  - Hôpitaux Universitaires La Pitié Salpêtrière-Charles Foix, Paris
  - Institut Curie, Paris
  - CHU Poitiers, Poitiers
  - CHU de Reims - American Memorial Hospital 2, Reims
  - Centre Eugène Marquis, Rennes
  - CHU Rennes - Hôpital Sud, Rennes
  - CHU Rouen Normandie - Hôpital Charles-Nicolle, Rouen
  - CHU de Saint-Denis de La Réunion, Saint-Denis
  - CHU de Saint-Etienne - Hôpital Nord, Saint-Etienne
  - CHU de Saint-Pierre de La Réunion Sud, Saint-Pierre
  - Centre Régional Lutte Contre le Cancer Paul STRAUSS, Strasbourg
  - Hôpital de Hautepierre, Strasbourg
  - Hôpital Foch, Suresnes
  - Hôpital des enfants, Toulouse
  - Institut Universitaire du Cancer de Toulouse-Oncopole (IUCT-O) - Institut Claudius Regaud, Toulouse
  - CHRU Tours - Hôpital Clocheville, Tours
  - CHRU Tours - Hôpital Bretonneau, Tours
- Spain (3):
  - Hospital Vall D´Hebron, Barcelona
  - Hospital Universitario Niño Jesus, Madrid
  - Hospital Universitario y Politécnico de La Fe, Valencia
- Karolinska University Hospital, Stockholm, Sweden